CLINICAL TRIAL: NCT01635491
Title: Gastrointestinal Transit Times and Motility in Healthy Volunteers Obtained by Motilis-3D-transit
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Motilis,Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: M-20100267
Record Dates: First submitted 2012-06-26; First posted 2012-07-09 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Gastrointestinal Motility; Total Gastrointestinal Transit Time; Segmental Transit Time; Gastric Emptying
Keywords: Gastrointestinal Motility; Transit time

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe gastrointestinal motility and transit times in healthy subjects by using Motilis 3D-Transit and to compare the total gastrointestinal transit time (GITT) to GITT obtained using radioopaque markers.

The investigators end points are to measure the transit times through different segments of the gastrointestinal canal,e.g. gastric emptying, small intestine, total GITT.

The study is descriptive and is designed to test and evaluate the usefulness of the Motilis 3D-Transit system. The investigators hypothesize, that with the system transit times through different segments of the gastrointestinal canal can be measured.

The design is made for evaluating the transit times, the inter-subject reproducibility and comparison with gold standard for colonic transit time measurement.

The investigators have chosen to include 20 healthy volunteers.The study is descriptive and therefore power calculation is not needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer
* Signed informed consent obtained
* Fasted since midnight

Exclusion Criteria:

* Subject has known GI related symptoms complaints or GI diseases, including swallowing disorders
* Subject has cancer or other life threatening diseases or conditions
* Subject is pregnant
* Subject has undergone abdominal surgery
* Subject has abdominal diameter >140cm?
* Drug abuse or alcoholism
* Subject's bowel movements are irregular
* Subject has known cardiovascular or pulmonary diseases
* Participation in any clinical study within the last 30 days
* Subject has cardiac pacemaker or infusion pump or any other implanted or portable electro-mechanical medical device.
* Subject takes any medication affecting GI motility
* Subject having MRI within the next four weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Total gastrointestinal transit time in healthy subjects. | Three days from baseline visit

SECONDARY OUTCOMES:
Segmental transit times in healthy subjects | Three days from Baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: AnneMette Haase, Ph.D Student, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Hepato and Gastroenterolegy, Aarhus, Denmark